CLINICAL TRIAL: NCT05987358
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Study to Evaluate the Efficacy and Safety of TQB3454 Tablets in the Treatment of Advanced Biliary Tract Cancer With Isocitrate Dehydrogenase 1 (IDH1) Mutation.
Brief Title: A Clinical Study of TQB3454 Tablets in the Treatment of Advanced Biliary Carcinoma.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB3454-III-01
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-03

CONDITIONS: Biliary Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3454 tablets (Experimental): TQB3454 tablets orally administered, 21 days as a treatment cycle.
  Interventions: Drug: TQB3454 tablets
- Placebo (Placebo Comparator): Placebo tablets orally administered, 21 days as a treatment cycle.
  Interventions: Drug: TQB3454 tablets matching placebo

INTERVENTIONS:
Drug: TQB3454 tablets — TQB3454 is a selective IDH1 mutant enzyme inhibitor.
  Arms: TQB3454 tablets
Drug: TQB3454 tablets matching placebo — Placebo tablets without active substance.
  Arms: Placebo

SUMMARY:
This study used a randomized, controlled, double-blind, multicenter Phase III clinical design with overall survival (OS) as the primary endpoint. About 165 patients with advanced biliary carcinoma were enrolled and randomly assigned to the experimental group and the control group in a 2:1 ratio to receive TQB3454 tablets or the placebo, respectively, to evaluate the efficacy and safety of TQB3454 tablets in the treatment of advanced biliary carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old, ≤75 years old (calculated on the date of signing the informed consent); Eastern Cooperative oncology Group (ECOG) score 0 ~ 2.
* Tumor tissue samples must be provided for genetic testing (10 puncture paraffin sections or 5 surgical paraffin sections).
* Patients with viral hepatitis: Patients should be treated symptomatically until the virus is stable before enrollment, and treatment should be maintained during the experimental period.
* The main organs have good functions.
* Meet the criteria for advanced biliary carcinoma:

  1. cholangiocarcinoma histologically or cytologically confirmed
  2. Locally advanced, relapsing, and/or metastatic disease that is not operable and has at least one measurable lesion according to Response Evaluation Criteria In Solid Tumors V1.1 (RECIST 1.1) criteria.
  3. Previous gemcitabine and fluorouracil (and/or platinum-based) drug therapy failed.
* Women of reproductive age should agree that they must use effective contraception during the study period and for 6 months after the study, and that serum or urine pregnancy tests are negative within 7 days prior to study enrollment; Men should agree that effective birth control must be used during the study period and for six months after the end of the study period.
* The subjects voluntarily joined the study, signed the informed consent, and the compliance was good.

Exclusion Criteria:

* Complicated diseases and medical history.

  1. The patient had or was currently present with other malignant tumors within 3 years prior to the first medication.
  2. Unmitigated toxic reactions above class 1 of Common Terminology Criteria for Adverse Events V5.0 (CTCAE) due to any previous treatment, excluding hair loss;
  3. Received major surgical treatment, significant traumatic injury, or long-standing unhealed wounds or fractures within 4 weeks prior to initial medication;
  4. Patients with any bleeding or bleeding events ≥CTCAE grade 3 within 4 weeks prior to initial administration; Patients with arteriovenous thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis and pulmonary embolism, occurring within 6 months prior to initial administration; Treatment with low molecular weight heparin was allowed and antiplatelet drugs were prohibited throughout the study;
  5. There is a history of active tuberculosis, idiopathic pulmonary fibrosis, institutional pneumonia, drug-induced pneumonia, radiation pneumonia requiring treatment or active pneumonia with clinical symptoms;
  6. Those who have the history of psychotropic drug abuse and cannot abstain or have mental disorders;
  7. Those who plan to undergo or have previously received allogeneic bone marrow transplantation or solid organ transplantation;
  8. A history of hepatic encephalopathy;
  9. Current or recent use (within 7 days prior to the start of study treatment) of aspirin (>325 mg/ day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel, and cilostazol;
  10. Subjects with any severe and/or uncontrolled medical conditions, including:

      1. Poor blood pressure control (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg);
      2. have grade 2 myocardial ischemia or myocardial infarction, arrhythmias (including Corrected Q-T interval (QTC) ≥ 450ms in men and 470ms in women), and grade 2 congestive heart failure (New York Heart Association (NYHA) rating);
      3. Active or uncontrolled severe infection (≥CTCAE grade 2 infection);
      4. Patients with renal failure requiring hemodialysis or peritoneal dialysis;
      5. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases;
      6. People who have epilepsy and need treatment.
* Tumor related and treatment:

  1. Hepatocellular carcinoma, fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, etc. confirmed by histology or cytology;
  2. According to imaging examination, cancer thrombus of the portal vein involved both the main trunk and the left and right primary branches, or involved both the main trunk and above veins (superior mesenteric vein, inferior mesenteric vein, spleen vein), or had cancer thrombus of the inferior vena cava or involved the heart;
  3. Uncontrolled pleural effusion, pericardial effusion or moderate to severe ascites that still require repeated drainage (the investigator's judgment);
  4. Known spinal cord compression, cancerous meningitis, symptoms of brain metastases, or symptoms controlled for less than 4 weeks.
* Research and treatment related:

  1. Known allergy to study drug excipients.
  2. Patients with multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
  3. Patients who require immunosuppressive, systemic, or absorbable topical hormone therapy for immunosuppressive purposes and who continue to use it within 7 days prior to initial administration (except for those whose daily dose of corticosteroids is less than 10 mg prednisone or other therapeutic hormones).
* Patients who participated in and used other antitumor clinical trials within 4 weeks before the first drug administration;
* According to the judgment of the researcher, there is any situation that seriously endangers the safety of the subject or affects the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 18 months.
  It refers to the time from randomization to the death from any cause.

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) | Up to 12 months.
  It refers to the time from randomization to disease progression or death, whichever occurs first.
Progression-Free-Survival 2 (PFS2) | Up to 3 months.
  The time between the first disease progression and the second disease progression or death, whichever comes first.
Objective Response Rate (ORR) | Up to 18 months.
  The percentage of subjects with complete response (CR) or partial response (PR).
Disease Control Rate (DCR) | Up to 18 months.
  The percentage of subjects with complete response (CR), partial response (PR) and stable disease (SD).
Duration of response (DOR) | Up to 7 months.
  The time from randomization to initiation of a new antitumor therapy or early termination of therapy.
The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) | Up to 18 months.
  It is an integrated system to describe the quality of life of cancer patients.
The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-BIL21) | Up to 18 months.
  It is an integrated system to describe the quality of life of cancer patients.
Incidence of adverse events (AE) | Up to 20 months.
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs) as assessed by Common Terminology Criteria for Adverse Events V5.0 (CTCAE 5.0)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Tangshan People's Hospital, Tangshan, Hebei
  - Third Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality